CLINICAL TRIAL: NCT02576886
Title: Combined Supine/Prone Acquisitions in Stress-First/Stress-Only Myocardial Perfusion Imaging to Reduce Equivocal Results in Patients Undergoing Testing in a Tertiary Care Facility
Brief Title: Combined Supine/Prone Acquisitions in Stress-First/Stress-Only Myocardial Perfusion Imaging to Reduce Equivocal Results
Acronym: SFSO-MPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 01-15-CARD-001
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Coronary Artery Disease
Keywords: supine; prone; myocardial perfusion imaging; radiation exposure; pre-screening tool
MeSH Terms: conditions — Coronary Artery Disease; Deception | interventions — Gamma Cameras

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Supine/Prone Imaging (Experimental): The patient will be imaged in the standard supine position and then an additional image will be acquired of the patient in the prone position.
  Interventions: Device: Gamma Camera; Procedure: Prone Imaging

INTERVENTIONS:
Device: Gamma Camera — All images acquired with the General Electric Discovery 530c
  Other Names: General Electric Discovery 530c
Procedure: Prone Imaging

SUMMARY:
Participants are being asked to participate in this research study because the participant's doctor has ordered a myocardial perfusion SPECT (Single-Photon Emission Computed Tomography) scan to look at the blood flow in the participants heart.

Myocardial perfusion imaging is a proven test that looks at the blood flow to the participant's heart after the injection of a radioactive tracer. The standard test requires two injections of the radioactive tracer and takes images of the participant's heart at rest and after a stress test. It has been proposed that in some cases, patients could have images done only after the stress portion of the test and, if normal, the rest images would not need to be done. In this case, only one injection of the radioactive tracer would be needed. It has further been proposed that adding another stress image made with the participant lying on their stomach, will increase the confidence of the reporting doctor in reporting stress images.

The purpose of this study is to find out if the extra information added from the image with the participant on their stomach helps the doctor when reporting the test results.

DETAILED DESCRIPTION:
Successfully implementing a SFSO-MPI protocol requires a validated pre-screening tool and a proven imaging protocol that aids the physician in reporting the study with confidence. The investigator's previous study, entitled "The feasibility of Stress-First/Stress-Only Myocardial Perfusion Imaging to reduce patient radiation exposure in a selected subset of patients undergoing testing in a tertiary care facility (SFSO-MPI)", was designed to validate a pre-screening tool developed by Duvall et al. In the investigator's population the tool demonstrated sensitivity and specificity (95% CI) of 0.79 (0.74-0.83) and 0.55 (0.48-0.62) (unpublished data). The sensitivity was lower than previous published. However the investigators noted that a greater proportion of participants were classified as abnormal (55% vs 31 and 36% in the two cohorts described by Duvall et al) and a high number of patients (15%) were reported as having equivocal stress images. These factors may have affected the sensitivity of the pre-screening tool. A greater proportion of the investigator's participants would then have required a rest study for proper interpretation of the test. Additional imaging increases the patients' radiation exposure and time requirement for the study and affects the proper allocation of department resources.

The department routinely images patients in only the supine position. The implementation of routine combined supine/prone imaging is expected to decrease image artifacts which may reduce the number of studies reported as equivocal. If combined supine/prone imaging is successful in changing the interpretation of a significant proportion of equivocal stress studies to normal, then the need for rest imaging will be obviated in a larger group of patients, resulting in reduced radiation dose to patients and medical staff, better laboratory efficiency due to faster throughput, reduced time commitment for patients and lower radiopharmaceutical cost. This change to practice will also further aid meeting the American Society of Nuclear Cardiology (ASNC) goal of no more than 9mSv patient exposure in 50% of studies.

ELIGIBILITY:
Inclusion Criteria:

* Any patient referred for a clinically indicated rest/stress myocardial perfusion imaging test

Exclusion Criteria:

* None

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Performance of the screening tool for each imaging protocol will be evaluated in terms of sensitivity and specificity to predict an unsuccessful SFSO study. | day of test
  The performance of the screening tool with supine-only and combined supine-prone imaging will be compared with a McNemar Chi-squared test for each of Group 1 and Group 2 to determine if the combined imaging protocol reduces equivocal results.

SECONDARY OUTCOMES:
Negative predictive value (i.e. the likelihood of successfully predicting a normal MPI based on the screening tool and a normal stress test) will be calculated for each of Group 1 and Group 2 with supine, and supine/prone imaging. | day of test
  The results for each group will be compared using a paired t-test, while results across groups will be compared using an unpaired t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Gulenchyn, MD,FRCPC, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton Health Sciences - Hamilton General Site, Hamilton, Ontario, Canada